CLINICAL TRIAL: NCT05355116
Title: A Comparison of Skin Temperature Changes Around the Knee When Using Cryocompression Devices
Brief Title: Different Cryocompression Devices and Skin Temperature of the Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Winchester (Other)
Collaborators: Physiolab Technologies Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HWB_REC_ 220228_Faulkner
Record Dates: First submitted 2022-03-24; First posted 2022-05-02 (Actual); Results first posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-10

CONDITIONS: Temperature Change, Body
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (5):
- Group A: Physiolab S1 (Experimental): The cryocompression device will be attached to the lower limb of participants using a cuff spanning from the mid-thigh to mid-calf. The device will exert an intermittent pressure of 25-50 mmHg throughout each test session. The device will pump temperature-controlled cold water through the cuff in order to reduce the skin temperature around the knee (and intra-articular temperature). The temperature of the water being pumped through the device will be 8℃. Each test session will last for 30 minutes. Participants will take part in all conditions, with at least 24 hours rest in between test sessions. Skin temperature around the knee will be measured prior to the cryocompression device being applied; every 5 minutes during the 30 minute test; and every 5 minutes after the test until skin temperature >15℃.
  Interventions: Device: Physiolab S1
- Group B: Breg Vpulse (Experimental): The cryocompression device will be attached to the lower limb of participants using a cuff spanning from the mid-thigh to mid-calf. The device will exert a dynamic peak pressure of 50 mmHg throughout each test session. The device will pump temperature-controlled cold water through the cuff in order to reduce the skin temperature around the knee (and intra-articular temperature). The temperature of the water being pumped through the device will not be lower than 5.5℃. The selected pressure and temperature represents the maximum capability of this device. Each test session will last for 30 minutes. Participants will take part in all conditions, with at least 24 hours rest in between test sessions. Skin temperature around the knee will be measured prior to the cryocompression device being applied; every 5 minutes during the 30 minute test; and every 5 minutes after the test until skin temperature >15℃.
  Interventions: Device: Breg Vpulse
- Group C: Cryo/Cuff (Experimental): The cryocompression device will be attached to the lower limb of participants using a cuff spanning from the mid-thigh to mid-calf. The pressure and temperature that the device applies to the treatment area is non-modifiable and undefined. The device will be used according to the manufacturer's recommendations, which will represent the maximum capability of this device. Each test session will last for 30 minutes. Participants will take part in all conditions, with at least 24 hours rest in between test sessions. Skin temperature around the knee will be measured prior to the cryocompression device being applied; every 5 minutes during the 30 minute test; and every 5 minutes after the test until skin temperature >15℃.
  Interventions: Device: Aircast Cryo/Cuff
- Group D: GameReady (Experimental): The cryocompression device will be attached to the lower limb of participants using a cuff spanning from the mid-thigh to mid-calf. The device will exert an intermittent pressure of 5-50 mmHg throughout each test session. The device will pump temperature-controlled cold water through the cuff in order to reduce the skin temperature around the knee (and intra-articular temperature). The temperature of the water being pumped through the device will be 1℃. Each test session will last for 30 minutes. Participants will take part in all conditions, with at least 24 hours rest in between test sessions. Skin temperature around the knee will be measured prior to the cryocompression device being applied; every 5 minutes during the 30 minute test; and every 5 minutes after the test until skin temperature >15℃.
  Interventions: Device: GameReady
- Group E: Physiolab Gel Therapy Wrap (Experimental): The cryocompression device will be attached to the lower limb of participants using a cuff spanning from the mid-thigh to mid-calf. The pressure and temperature that the device applies to the treatment area is non-modifiable and undefined. The device will be used according to the manufacturer's recommendations, which will represent the maximum capability of this device. Each test session will last for 30 minutes. Participants will take part in all conditions, with at least 24 hours rest in between test sessions. Skin temperature around the knee will be measured prior to the cryocompression device being applied; every 5 minutes during the 30 minute test; and every 5 minutes after the test until skin temperature >15℃.
  Interventions: Device: Physiolab Gel Therapy Wrap

INTERVENTIONS:
Device: Physiolab S1 — A cryocompression device capable of circulating ice-water through a cuff at 6-12℃ with either a static pressure of 25mmHg or dynamic pressure of 25-50 mmHg or 25-75mmHg. The lowest temperature setting, and highest pressure setting will be used for this study.
  Arms: Group A: Physiolab S1
Device: Breg Vpulse — A cryocompression device capable of circulating ice-water through a cuff at no lower than 5.5℃ with a dynamic peak pressure of 50 mmHg. The temperature of the ice-water, and the applied pressure, is not modifiable by the user.
  Arms: Group B: Breg Vpulse
Device: Aircast Cryo/Cuff — A cryocompression device capable of circulating ice-water through a cuff at an undefined, non-modifiable temperature with a static pressure that is also undefined and non-modifiable. The device will be applied as per the manufacturer's instructions, which will represent its maximum capability.
  Arms: Group C: Cryo/Cuff
Device: GameReady — A cryocompression device capable of circulating ice-water through a cuff at 1-12℃ with a dynamic pressure of 5-15 mmHg, 5-50 mmHg, or 5-75 mmHg. The lowest temperature setting, and highest pressure setting will be used for this study.
  Arms: Group D: GameReady
Device: Physiolab Gel Therapy Wrap — A cryocompression cuff that applies an undefined, non-modifiable temperature with a static pressure that is also undefined and non-modifiable. The device will be applied as per the manufacturer's instructions, which will represent its maximum capability.
  Arms: Group E: Physiolab Gel Therapy Wrap

SUMMARY:
Cryotherapy after surgery is widely utilised and has numerous practical applications for post-operative rehabilitation. Previous research has suggested that during cold therapy, the skin temperature of the knee should be reduced to 10-15°C to maximise the therapeutic benefits of cooling while avoiding the risk of cold injuries such as nerve damage and frostbite (Wilke and Weiner, 2003; Bleakley, McDonough and MacAuley, 2004). However, a recent study noted that where cryocompression devices have previously been used to reduce the skin temperature <10°C, no complications relating to the device have been reported, suggesting that the risk to the user at these lower temperatures is minimal (Bellon et al., 2019). The temperature range at which a cryocompression device should be set in order to achieve a skin temperature within the therapeutic range of 10-15°C is unknown. Furthermore, there is evidence to suggest that the temperature setting of the device does not equal that to which the skin is reduced (Selfe et al., 2009). Therefore, it is not sufficient to assume that the temperature setting of a cryocompression device accurately reflects skin temperature. Modern cryotherapy devices often consist of some sort of cuff that can be wrapped around the knee, with a connecting tube to a central unit that supplies and circulates ice-water to and from the cuff in order to cool the intended body part. Such devices offer differing levels of control over the temperature of the ice-water as it leaves the central unit, but nothing is known about how this correlates to the skin temperatures that are achieved during a cryotherapy treatment.

The aim of this study is to determine the ability of five different cryocompression.devices to effectively lower the skin temperature of the treatment area to within the therapeutic range.

DETAILED DESCRIPTION:
Design This prospective randomised controlled trial will recruit healthy adult volunteers from a university population to participate. A power analysis demonstrated that a total of 30 participants would be required to achieve a power of 0.8 and alpha error probability of 0.05 for a small-medium effect size of f=0.2. Each participant will take part in every condition to eliminate the risk of demographic factors confounding the results. Each of the 5 devices being investigated will comprise each of the test conditions. The order in which participants complete the 5 test conditions will be randomised in advance using a computer random number generator. Testing will involve each device being applied and used according to the manufacturers' recommendations. Each testing session will take around 60 minutes to complete, depending on the treatment application guidelines of each device, with at least 24 hours between tests involving the same participant. In total, participants will be giving around 5 hours of time across 5 days to complete their participation.

Protocol All eligible participants will first be required to provide informed consent prior to their participation in the study. Once this has been obtained, participants will each attend 5 individual testing sessions, each lasting no longer than 60 minutes. The height and mass of the participants will be measured during the first testing session in order to calculate BMI, and participants' age and sex will be recorded and included in the later data analysis.

Participants will be required to remain in a seated position with their leg in full extension and elevated, parallel to the floor, for the duration of each test. The leg that will be used for the study will be randomly selected for each participant, and will remain the same for each condition. Skin temperature will be measured using a thermocouple, which will be attached with tape 20 mm distal to the patella. One of the cryocompression devices (Physiolab S1; Physiolab ice pack; GameReady; Cryo/Cuff; or VPulse) will then be attached to the leg of the participant and the test will begin. Depending on the condition to which a participant has been randomly assigned for a given test, a different device will be used. The temperature and pressure settings for each test will be set according to the maximum capability of each device, which varies between devices. The lowest temperature setting that will be used throughout the study will be 1℃ (GameReady device) and the highest pressure setting that will be used is 50 mmHg (GameReady and Physiolab S1 devices). None of the temperature or pressure settings used are deemed to be unsafe or have a high risk of adverse reactions, as long as participants are not contraindicated according to the exclusion criteria for this study.

The temperature of the skin will be measured using a k-type thermocouple attached to an infrared thermometer immediately prior to the application of a device, and then every 5 minutes for the duration of the test. The length of a test will be 30 minutes, in accordance with the manufacturers' instructions/recommendations for each device.

Upon completion of a test, the cuff will be removed. If the temperature of the skin has been reduced to within 10-15℃, skin temperature will continue to be monitored every 5 minutes after the cuff has been removed until it rises above 15℃, at which point the test will end. This will allow for the total time to be measured that skin temperature remains within the target therapeutic range as a result of a single application of the cryocompression device. If the skin temperature is not reduced to within 10-15℃ while the cuff is worn, then the test will end after the cuff is initially removed. Upon completion of the test, the temperature sensor will be removed from the leg of the participant; thus completing their participation in the test. Once each participant has taken part in all conditions, they will have completed their participation in the study.

The following measures will be recorded: skin temperature at each time point, minimum skin temperature achieved, time to achieve minimum skin temperature, length of time with skin temperature within therapeutic range of 10-15℃. After each test, participants will also be asked to respond to the following question using a 5-point Likert scale: "How comfortable did you find the treatment you just experienced?" The possible answers to this question will be: "Very comfortable, Comfortable, Neutral, Uncomfortable, Very uncomfortable". This will provide insight into differences in perception of the treatment, which could be relevant for the likelihood of protocol adherence by patients in clinical settings.

Analysis The data will be analysed to detect any differences during testing compared to baseline measures, and between groups. All data will be first subjected to a Kolmogorov-Smirnov test to assess whether they are normally distributed. A repeated measures analysis of variance will be performed on all normally distributed data. A Friedman test will be performed on any data that are not normally distributed.

Ethical issues There is a low risk of cold injury to participants if their skin temperature is reduced to <10℃ for any prolonged period of time (>60 mins). The coldest temperature setting for this study is 1℃ (GameReady), which will be applied for 30 mins. However, device temperature settings do not equal the actual skin temperatures achieved, and it is not expected that skin temperatures will be reduced to lower than 5℃ for more than 15 minutes during any test. Therefore, the risk of harm to the participant is deemed to be minimal for this study.

Participants have the right to withdraw themselves and any collected data from the study at any time during, and for the first 7 days after, their participation without having to give a reason. They also have the right to terminate a test session at any time. Testing shall also be terminated as a result of any adverse reactions that emerge. Adverse reactions (e.g. pain) to the testing protocol are not expected due to the low-risk nature of the study, however any that occur shall be recorded and monitored until things return to baseline/normal. In order to monitor any pain/discomfort that might occur, a Numerical Pain Rating Scale (0-10 scale) will be within sight of the participant at all times during testing: a test will be terminated if reported pain/discomfort exceeds 5/10, though none is expected. Any reported pain (or other adverse reactions) shall be stored along with the data collected for that participant. If a test is terminated for a reason that could be mitigated in future, participants will be offered the opportunity to repeat the test another day, should they wish to continue taking part in the study. If a test is terminated due to an adverse reaction that can not be mitigated in future, the participant (and any collect-ed data) will be thanked for their time and withdrawn from the study.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age

Exclusion Criteria:

* • BMI >40 kg/m2

  * History of nerve damage or sensory deficit in the lower limbs (including frostbite)
  * Hypersensitivity to cold, including hives
  * Active inflammation or pain of the knee
  * History of thrombosis, embolism, or other conditions related to impaired peripheral circulation
  * Suffering from diagnosed diabetes, multiple sclerosis, rheumatoid arthritis, spinal cord injury, cardio-vascular disease, hypertension, Raynaud disease, cryoglobulinemia, or haemoglobinuria
  * Confirmed or suspected tissue infection, an unstable fracture, a skin condition, or a tumour in the treatment area
  * Cognitive impairment or communication barriers where adjustments can not be reasonably made

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Faulkner, PhD, Principal Investigator — University of Winchester
Locations (1):
- Physiology Laboratory, Winchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual data will be shared outside of the researchers directly involved in the data collection itself.

REFERENCES:
- [Background] Wilke B, Weiner RD. Postoperative cryotherapy: risks versus benefits of continuous-flow cryotherapy units. Clin Podiatr Med Surg. 2003 Apr;20(2):307-22. doi: 10.1016/S0891-8422(03)00009-0. PMID 12776983
- [Background] Bleakley C, McDonough S, MacAuley D. The use of ice in the treatment of acute soft-tissue injury: a systematic review of randomized controlled trials. Am J Sports Med. 2004 Jan-Feb;32(1):251-61. doi: 10.1177/0363546503260757. PMID 14754753
- [Background] Fang L, Hung CH, Wu SL, Fang SH, Stocker J. The effects of cryotherapy in relieving postarthroscopy pain. J Clin Nurs. 2012 Mar;21(5-6):636-43. doi: 10.1111/j.1365-2702.2010.03531.x. Epub 2011 Feb 20. PMID 21332855
- [Background] Waterman B, Walker JJ, Swaims C, Shortt M, Todd MS, Machen SM, Owens BD. The efficacy of combined cryotherapy and compression compared with cryotherapy alone following anterior cruciate ligament reconstruction. J Knee Surg. 2012 May;25(2):155-60. doi: 10.1055/s-0031-1299650. PMID 22928433
- [Background] Bellon M, Michelet D, Carrara N, Vacher T, Gafsou B, Ilhareborde B, Mazda K, Ferrero E, Simon AL, Julien-Marsollier F, Dahmani S. Efficacy of the Game Ready(R) cooling device on postoperative analgesia after scoliosis surgery in children. Eur Spine J. 2019 Jun;28(6):1257-1264. doi: 10.1007/s00586-019-05886-6. Epub 2019 Jan 31. PMID 30847706
- [Background] Selfe J, Hardaker N, Whittaker J and Hayes C. An investigation into the effect on skin surface temperature of three cryotherapy modalities. Thermology International. 2009; 19(4): 121-126.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adult participants were recruited from a University population between April 2022 and July 2022. The data collection took place in a University laboratory.
Pre-assignment Details: 32 participants were enrolled and began the data collection phase.
Groups:
- All Study Participants: This study employed a crossover design, wherein each of the participants received a 30-minute cryocompression treatment with all of the 5 modalities under investigation. The order in which each participation underwent a treatment with each modality was conducted in a randomised manner.
Period: Overall Study
Arm/Group | All Study Participants
Started (The number of participants enrolled to receive each treatment condition (in a randomised order)) | 32
Physiolab S1 (The number of participants who received a treatment with the Physiolab S1 device.) | 32
Breg VPulse (The number of participants who received a treatment with the Breg VPulse device) | 31
Cryo/Cuff (The number of participants who received a treatment with the Cryo/Cuff device.) | 31
GameReady (The number of participants who received a treatment with the GameReady device.) | 30
Gel Wrap (The number of participants who received a treatment with the Gel Wrap.) | 31
Completed (The number of participants who completed their participation in the study by receiving a treatment with each of the 5 devices under investigation.) | 30
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Although 32 participants were originally enrolled, only the data from 30 participants was included in the final analysis due to the withdrawal of 2 participants from the study for unknown reasons prior to their completion of all test conditions.
Groups:
- All Study Participants: According to a randomised order, each participant had the relevant cryocompression device attached to their lower limb using a cuff positioned centrally over the knee. Where relevant, each device was applied according to the manufacturer's guidelines, or where unclear, according to precedent in the literature. Each treatment lasted for 30 minutes. Participants took part in all conditions, with at least 24 hours rest in between test sessions. Skin temperature around the knee was measured prior to the cryocompression device being applied; every 5 minutes during the 30 minute test; and every 5 minutes after the test until skin temperature >15℃.
Arm/Group | All Study Participants
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.3 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 32
Leg (L:R) [Number; unit: Legs]
  Left | 16
  Right | 16
Height (m) [Mean (Standard Deviation); unit: metres] | 1.75 (0.1)
Mass (kg) [Mean (Standard Deviation); unit: kilograms] | 76.3 (10.1)
Body mass index (kg/m2) [Mean (Standard Deviation); unit: kilograms per square metre] | 24.8 (2.7)
Skin temperature (°C) [Mean (Standard Deviation); unit: degrees celsius] | 31.4 (1.8)
Ambient temperature (°C) [Mean (Standard Deviation); unit: degrees celsius] | 21.8 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Skin Temperature
Description: Skin temperature will be measured using a thermocouple positioned 20 mm distal to the patella. This sensor will be attached prior to the cryocompression device being applied, and will remain in place until the testing session is complete and skin temperature is >15℃. (The therapeutic skin temperature range for cryotherapy is thought to be 10-15℃). Temperature will be measured prior to the cryocompression device being applied; every 5 minutes during the test; and every 5 minutes after a test until the skin temperature reaches >15℃.
Time Frame: Up to 40 minutes per treatment
Population: Individuals who completed their participation in all test conditions were included in the final analysis.
Measure: Mean (Standard Deviation); unit: degrees celsius
Groups:
- Group A: Physiolab S1: The cryocompression device was attached to the lower limb of participants using a cuff spanning positioned centrally over the knee. The device exerted an intermittent pressure of 25-50 mmHg throughout each test session. The temperature of the water being pumped through the device was 8℃. Each treatment lasted for 30 minutes. The termperature and compression settings were chosen in line with the manufacturer recommendations. Participants took part in all conditions, with at least 24 hours rest in between test sessions. Skin temperature around the knee was measured prior to the cryocompression device being applied; every 5 minutes during the 30 minute test; and every 5 minutes after the test until skin temperature >15℃.
- Group B: Breg Vpulse: The cryocompression device was attached to the lower limb of participants using a cuff spanning positioned centrally over the knee. The device exerted the default level of intermittent compression throughout each test session. The temperature of the water pumped through the device was not lower than 5.5℃ and was not user-modifiable. Each test session lasted for 30 minutes. Participants took part in all conditions, with at least 24 hours rest in between test sessions. Skin temperature around the knee was measured prior to the cryocompression device being applied; every 5 minutes during the 30 minute test; and every 5 minutes after the test until skin temperature >15℃.
- Group C: Cryo/Cuff: The cryocompression device was attached to the lower limb of participants using a cuff spanning positioned centrally over the knee. The pressure and temperature that the device applied to the treatment area was non-modifiable and undefined. The device was used according to the manufacturer's recommendations. Each treatment lasted for 30 minutes. Participants took part in all conditions, with at least 24 hours rest in between test sessions. Skin temperature around the knee was measured prior to the cryocompression device being applied; every 5 minutes during the 30 minute test; and every 5 minutes after the test until skin temperature >15℃.
- Group D: GameReady: The cryocompression device was attached to the lower limb of participants using a cuff spanning positioned centrally over the knee. The device exerted an intermittent pressure of 5-50 mmHg throughout each test session, in line with manufacturer's recommendation. The temperature of the water pumped through the device was 1℃, in line with the precedent set in the literature and in lieu of a specific temperature setting recommended by the manufacturer. Each test session lasted for 30 minutes. Participants took part in all conditions, with at least 24 hours rest in between test sessions. Skin temperature around the knee was measured prior to the cryocompression device being applied; every 5 minutes during the 30 minute test; and every 5 minutes after the test until skin temperature >15℃.
- Group E: Physiolab Gel Therapy Wrap: The cryocompression device was attached to the lower limb of participants using a cuff spanning positioned centrally over the knee. The pressure and temperature that the device applied to the treatment area was non-modifiable and undefined. The device was used according to the manufacturer's recommendations. Each test session lasted for 30 minutes. Participants took part in all conditions, with at least 24 hours rest in between test sessions. Skin temperature around the knee was measured prior to the cryocompression device being applied; every 5 minutes during the 30 minute test; and every 5 minutes after the test until skin temperature >15℃.
Arm/Group | Group A: Physiolab S1 | Group B: Breg Vpulse | Group C: Cryo/Cuff | Group D: GameReady | Group E: Physiolab Gel Therapy Wrap
Number analyzed (Participants) | 30 | 30 | 30 | 30 | 30
degrees celsius
  Baseline skin temp | 31.18 (2.34) | 31.21 (1.46) | 31.1 (1.81) | 31.93 (1.8) | 31.39 (1.45)
  Skin temp after 5 mins | 19.97 (2.0) | 26.78 (3.17) | 24.15 (3.19) | 21.96 (2.95) | 21.2 (3.22)
  Skin temp after 10 mins | 18.2 (1.8) | 23.94 (2.89) | 21.92 (3.54) | 19.39 (2.9) | 20.22 (3.33)
  Skin temp after 15 mins | 16.08 (1.18) | 21.55 (2.89) | 20.39 (3.37) | 16.69 (2.59) | 19.58 (3.12)
  Skin temp after 20 mins | 15.12 (1.05) | 19.89 (3.2) | 18.92 (3.04) | 15.32 (2.1) | 19.48 (3.0)
  Skin temp after 25 mins | 14.52 (0.96) | 18.36 (2.72) | 18.31 (2.86) | 14.03 (1.85) | 19.6 (2.94)
  Skin temp after 30 mins | 13.94 (0.78) | 17.24 (2.64) | 17.01 (2.93) | 13.02 (1.64) | 19.86 (2.85)
  Skin temp after 35 mins: number analyzed (Participants) | 28 | 5 | 4 | 25 | 1
  Skin temp after 35 mins | 17.23 (2.18) | 21.62 (1.3) | 18.45 (2.49) | 17.96 (2.35) | 18.3 (NA) — Test had ended for all other participants except one prior to this time point due to skin temperature being >15 degrees Celsius. Since data only exist for a single participant at this time point, standard deviation is not relevant.
  Skin temp after 40 mins: number analyzed (Participants) | 3 | 0 | 0 | 2 | 0
  Skin temp after 40 mins | 19.07 (0.97) |  |  | 18.0 (0.57) |

2. Secondary Outcome: Subjective Comfort
Description: After each test, participants will also be asked to respond to the following question using a 5-point Likert scale: "How comfortable did you find the treatment you just experienced?" The possible answers to this ques-tion will be: "Very comfortable, Comfortable, Neutral, Uncomfortable, Very uncomfortable". This will provide insight into differences in perception of the treatment, which could be relevant for the likelihood of protocol adherence by patients in clinical settings.
Time Frame: 1 minute - recorded once immediately following treatments with each of the 5 devices under investigation
Population: Data were analysed for the 30 participants who fully completed their participation in the study.
Measure: Number; unit: percent
Arm/Group | Group A: Physiolab S1 | Group B: Breg Vpulse | Group C: Cryo/Cuff | Group D: GameReady | Group E: Physiolab Gel Therapy Wrap
Number analyzed (Participants) | 30 | 30 | 30 | 30 | 30
percent
  Participants reporting positive comfort ratings | 86.7 | 86.7 | 90.0 | 53.3 | 96.7
  Participants reporting neutral comfort ratings | 13.3 | 10.0 | 10.0 | 30.0 | 3.3
  Participants reporting negative comfort ratings | 0 | 3.3 | 0.0 | 16.7 | 0.0

ADVERSE EVENTS:
Time Frame: Each participant was monitored for adverse events during each test session, which was up to 60 minutes per treatment including arrival to the lab, testing, and post-test data collection/administration.
Description: There was deemed to be little-to-no risk of all-cause mortality or serious adverse events due to the screening process that occurred prior to participant enrollment. Only people who met the inclusion criteria and were not otherwise contraindicated for cryocompression therapy were able to participate.
Arm/Group | Group A: Physiolab S1 | Group B: Breg Vpulse | Group C: Cryo/Cuff | Group D: GameReady | Group E: Physiolab Gel Therapy Wrap
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32 | 0/32 | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/32 | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/32 | 0/32 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-11): https://cdn.clinicaltrials.gov/large-docs/16/NCT05355116/Prot_SAP_000.pdf